CLINICAL TRIAL: NCT02629653
Title: Body Cooling During Carotid Endarterectomy: No-profit, Open, Mono-centric, Feasibility Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: S. Andrea Hospital (Other)
Responsible Party: Principal Investigator, Francesco Orzi, Prof, MD, S. Andrea Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CEAC-0613
Record Dates: First submitted 2015-12-10; First posted 2015-12-14 (Estimated); Last update posted 2015-12-14 (Estimated); Status verified 2015-12

CONDITIONS: Carotid Artery Diseases; Hypothermia; Stroke; Carotid Artery Plaque; Carotid Artery Stenosis; Cerebrovascular Accident
Keywords: carotid endarterectomy; stroke; hypothermia; endovascular cooling
MeSH Terms: conditions — Carotid Artery Diseases; Hypothermia; Stroke; Carotid Stenosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Single arm (Other): The endovascular cooling system will be Zoll IVTM. This system consists of a control module (either CoolGard 3000 or Thermogard XP), a CoolGard start-up kit, and an ICY catheter (either IC-3585 AE or IC-3585)
  Interventions: Device: endovascular cooling (Zoll system)

INTERVENTIONS:
Device: endovascular cooling (Zoll system) — The Zoll IVTM is an endovascular cooling system that consists of a control module (either CoolGard 3000 or Thermogard XP), a CoolGard start-up kit, and an ICY catheter (either IC-3585 AE or IC-3585).

SUMMARY:
Aim of the study is to determine whether endovascular systemic cooling to a target temperature of 34-35°C initiated before, and maintained during Carotid EndoArterectomy (CEA), is feasible and safe

DETAILED DESCRIPTION:
The study is based on the hypothesis that performing CEA during hypothermia substantially reduces the risk due to a potential, temporary hypoperfusion, associated with the surgical procedure.

The rationale behind the study is based on the assumption that Carotid EndArterectomy (CEA), by removing local causes of downstream altered circulation, improves cerebral hemodynamics and provides an effective prevention of stroke and TIA. The intervention itself, however, causes immediate risk of stroke or death, and it is also an issue whether the temporary reduction of blood flow associated with clamping of the artery, during the surgical intervention, may trigger long-lasting brain tissue dysfunction.

Mild hypothermia (34-35 °C) is probably the most effective approach to protect the brain from ischemic insults. Most of the supportive data were obtained in animal models of ischemia. Several phase II trials have shown safety and feasibility of cooling subjects with stroke, in the hours following onset of symptoms. Early interventions show the highest benefit.

Eligible patients will initiate cooling 60-90 min before CEA with endovascular cooling (Zoll system) to the target 34-35°C (assessed by bladder thermometer). The Zoll IVTM system is an endovascular cooling system that consists of a control module (either CoolGard 3000 or Thermogard XP), a CoolGard start-up kit, an ICY catheter (either IC-3585 AE or IC-3585 CO or IC-3893 AE or IC-3893 CO), a catheter convenience kit for catheter insertion (CO models only), thermal probes and cables. All the devise component have CE mark. The Low temperature will be maintained during the CEA procedure, followed by gradual, passive, controlled rewarming (0.4 °C/h). Type of anaesthesia will be decided according to good clinical practice. The cooling procedure will be, therefore, carried out during the anaesthesia procedure required by the surgical intervention. There is a chance that the duration of the anaesthesia will be longer that required, but all the efforts will be undertaken to keep the anaesthesia time as short as if there were no cooling

Clinical and instrumental evaluations will be carried out before and post intervention. Each evaluation will consist of physical examination, neuropsychological evaluation (MoCA test), blood tests and brain MRI or TC.

Safety is evaluated on the basis of severe adverse event

ELIGIBILITY:
Inclusion Criteria:

1. Subject eligible for CEA, without progression of symptoms, with low (<4) Anesthesia Risk Assessment
2. Age ≥ 18 years;
3. Written informed consent

Exclusion Criteria:

1. Evidence from a CT or MRI scan or from other pre-inclusion investigations of an intracranial haemorrhage, a tumour, encephalitis, or any diagnosis of acute brain focal lesion;
2. Progression or instability of neurological status
3. Conditions that may be exacerbated by hypothermia, such as haematological dyscrasias, oral anticoagulant treatment with INR ≥ 1.7, severe pulmonary disease, severe heart failure (defined as a New York Heart Association (NYHA) score of III or IV), history of myocardial infarction within the previous 3 months, angina pectoris in the previous 3 months, severe infection with a C-reactive protein > 50 mg/dl, or a clinical diagnosis of sepsis;
4. Blood oxygen saturation below 94%, allowing a maximum of 2 L/min oxygen delivered nasally to achieve this;
5. Bradycardia (<40 beats/min);
6. Body weight > 120 kg;
7. Severe hepatic dysfunction, or severe renal dysfunction;
8. Pregnancy. Women of childbearing potential are excluded unless a negative test for pregnancy has been obtained prior to randomisation;
9. Other serious illness that may confound treatment assessment or increase the risks of cooling;
10. Social or other conditions that according to the investigator's judgement might be a major problem for follow-up.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2013-12; Primary Completion 2015-06 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Adverse events | Any adverse event at 1 month
  Severe adverse events were defined as any life-threatening event including pneumonia (diagnosed on the basis of clinical signs or symptoms), myocardial infarction and parenchymal hemorrhage. Non-severe safety outcomes included incidence of bradycardia (<40 beats per minute), cardiac arrhythmia, hypertension, hypotension and any coagulation disorders.

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Orzi, Prof, MD, Study Chair — NESMOS Department, University of Rome "La Sapienza"; St. Andrea Hospital
Locations (1):
- NESMOS Department St. Andrea Hospital, Rome, Rome, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Grotta JC. Clinical practice. Carotid stenosis. N Engl J Med. 2013 Sep 19;369(12):1143-50. doi: 10.1056/NEJMcp1214999. No abstract available. PMID 24047063
- [Result] Lee JH, Suh BY. Risk factor analysis of new brain lesions associated with carotid endarterectmy. Ann Surg Treat Res. 2014 Jan;86(1):39-44. doi: 10.4174/astr.2014.86.1.39. Epub 2014 Jan 1. PMID 24761406
- [Result] Endarterectomy for asymptomatic carotid artery stenosis. Executive Committee for the Asymptomatic Carotid Atherosclerosis Study. JAMA. 1995 May 10;273(18):1421-8. PMID 7723155
- [Result] Yenari MA, Han HS. Neuroprotective mechanisms of hypothermia in brain ischaemia. Nat Rev Neurosci. 2012 Feb 22;13(4):267-78. doi: 10.1038/nrn3174. PMID 22353781
- [Result] Erecinska M, Thoresen M, Silver IA. Effects of hypothermia on energy metabolism in Mammalian central nervous system. J Cereb Blood Flow Metab. 2003 May;23(5):513-30. doi: 10.1097/01.WCB.0000066287.21705.21. PMID 12771566
- [Result] Wu TC, Grotta JC. Hypothermia for acute ischaemic stroke. Lancet Neurol. 2013 Mar;12(3):275-84. doi: 10.1016/S1474-4422(13)70013-9. PMID 23415567
- [Result] van der Worp HB, Macleod MR, Kollmar R; European Stroke Research Network for Hypothermia (EuroHYP). Therapeutic hypothermia for acute ischemic stroke: ready to start large randomized trials? J Cereb Blood Flow Metab. 2010 Jun;30(6):1079-93. doi: 10.1038/jcbfm.2010.44. Epub 2010 Mar 31. PMID 20354545
- [Result] Kamme F, Campbell K, Wieloch T. Biphasic expression of the fos and jun families of transcription factors following transient forebrain ischaemia in the rat. Effect of hypothermia. Eur J Neurosci. 1995 Oct 1;7(10):2007-16. doi: 10.1111/j.1460-9568.1995.tb00623.x. PMID 8542058
- [Derived] Candela S, Dito R, Casolla B, Silvestri E, Sette G, Filippi F, Taurino M, Brancadoro D, Orzi F. Hypothermia during Carotid Endarterectomy: A Safety Study. PLoS One. 2016 Apr 8;11(4):e0152658. doi: 10.1371/journal.pone.0152658. eCollection 2016. PMID 27058874